CLINICAL TRIAL: NCT04253665
Title: Nursing Discharge Teaching for Multimorbid Inpatients to Self-manage Their Health at Home: a Pilot Study
Brief Title: Nursing Discharge Teaching for Multimorbid Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Dr. Sc. Cedric Mabire, RN PhD, Dr.Sc., University of Lausanne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020_2201
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Chronic Disease
Keywords: Discharge teaching; Nursing; Multimorbidity
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: 2 group pre/post-intervention comparative design: 90 control patients will be recruited before the implementation of the intervention in study units. This recruitment will last approximately two months, according to the estimated turnout of patients in these units. After this control period, 30 other patients will be recruited to receive the intervention. In this sense, participants are assigned to one group or the other, depending on the phase of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Discharge teaching is usually not delivered in a systematic or consistenly way, nor by relying on a particular intervention model.
- Discharge teaching (Experimental): Receiving tailored discharge teaching by nurses during hospital stay.
  Interventions: Behavioral: Nursing discharge teaching

INTERVENTIONS:
Behavioral: Nursing discharge teaching — Nurses will provide multimorbid seniors inpatients with teaching related to self-management to prepare them to be discharged home. The teaching delivery will be tailored to patients' activation level and priorities. The intervention begins by determining the level of activation at which patients are and identifying priorities to address related to patients' life situation. A Discharge Teaching Guide will be used by nurses to deliver the teaching and includes six domains of self-management. For each domain, nurses first report whether a priority has been identified and what intervention they have proposed to address it. Then for each domain, teaching objectives are described and differ according to the level of patient activation. These six domains of self-management are found in the patient-oriented discharge summary, which is a document for the patient that summarizes what has been addressed in discharge teaching.
  Arms: Discharge teaching

SUMMARY:
The objective of this study is to estimate the effect size of a nursing discharge teaching intervention on multimorbid inpatients activation level, health confidence, readiness for hospital discharge, experience with discharge care and rate and time to 7-days readmission.

DETAILED DESCRIPTION:
Seniors returning home from hospital have to manage several chronic conditions in addition to their daily tasks. The teaching provided by nurses during hospitalization is essential care to prepare them to manage their health at home. Nevertheless, there is often a gap between professionals' belief that the teaching they have provided to patients has met their needs, and patients' perceptions of the relevance of the teaching content to their home situation. The time available to conduct this teaching is also short during the hospital stay and there is limited knowledge about how to adapt this teaching for patients who must manage multiple chronic conditions at the same time. Thus, there is a real need to develop and test a new teaching nursing intervention to prepare for the return home that takes into account the unique and complex needs and characteristics of patients with multiple chronic conditions. Tailoring teaching to seniors' life situation and level of activation (i.e., knowledge, skills and confidence in managing their health) would best meet the needs of these patients for managing their health at home. An intervention that takes these characteristics into account has been developed and will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* 2 chronic diseases or more
* Being discharged home
* Able to speak, read and write in French

Exclusion Criteria:

* Insufficient capacity to consent assessed with the University of California San Diego Brief Assessment of Capacity to Consent (UBACC).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Activation Measure (PAM) | change from hospital admission to the day of discharge and 7-10 days after discharge
  The patient activation measure (PAM) is a 13-item self-report questionnaire to measure patient activation level. Stages of activation are distributed as follows in the PAM items: items 1-2: believing an active role is important; items 3-8: having confidence and knowledge to take action; items 9-11: taking action; and items 12-13: continuing healthy behaviors under stress. PAM raw score can be calculated by adding all of the responses to the 13 questions. This score is then converted into an activation score ranging from 0 = no activation to 100 = high activation using a calibration table. Psychometric properties of the PAM in hospitalized multimorbid patients showed a satisfying reliability (Cronbach's alpha = 0.88) and a content validity index of 0.91.

SECONDARY OUTCOMES:
Change in Health Confidence Score (HCS) | change from hospital admission to the day of discharge and 7-10 days after discharge
  The Health Confidence Score (HCS) is an easy-to-obtain proxy measure for the patient activation construct. The HCS is a short measure (4-items) of patients' confidence to manage their health and engage with healthcare providers. Four dimensions are explored: Knowledge, Self-management, Access to help, Shared decision-making. Items have four response options (3 = strongly agree, 2 = agree, 1 = neutral, 0 = disagree). Scores are reported for each item and the higher they are, the higher the confidence is. A summary score is calculated with a 13-point scale by adding the individual items scores, with a range from 0 (4×disagree) to the ceiling 12 (4×strongly agree). This instrument has good internal consistency (Cronbach's alpha = 0.82) and construct validity.
Readiness for Hospital Discharge Scale-Short Form (RHDS-SF) | At the end of the hospital stay, an average of 7-10 days after admission
  Readiness for hospital discharge is an estimate by the patient of having the ability to leave the hospital, to be ready to face the realities of everyday life at home and the needs generated by their new health condition. The Readiness for Hospital Discharge Scale-Short Form (RHDS-SF) is an eight items self-reported questionnaire. Four dimensions measure personal status, knowledge to manage the post-hospital period, the ability to adapt to new health needs and the expected support. Each item is scored on a Likert scale from 0 to 10, with the highest score indicating a better perceived readiness. A mean score greater than or equal to 7 indicates that the patient is ready for hospital discharge. Content and construct validity of the RHDS-SF are missing so far. Predictive validity was tested but results showed that the patient short form of the RHDS cannot predict 30-day readmissions and emergency department visits. The RHDS has a Cronbach's alpha of 0.79.
Readmission rate and time to readmission | 7-10 days after discharge
  7-10-day readmission rate and time to readmission retrieved from medical charts
Discharge Care Experiences Survey (DICARES) | 7-10 days after discharge
  This 11-items instrument investigates three domains: coping after discharge (4 items), adherence to treatment (3 items) and participation in discharge planning (4 items). The answer for each item ranges from 1 ("Not at all") to 5 ("To a very large extent"), with higher scores indicating more positive experience. The psychometric evaluation of the DICARES in senior patients showed an excellent test-retest reliability (ICC = 0.76, CI 95%[0.70, 0.82]), satisfactory construct validity (r = 0.54, p <0.01) and an acceptable internal consistency (Cronbach's alpha = 0.82).

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Mabire, Dr. Sc., Principal Investigator — Institute of Higher Education and Research in Healthcare, University of Lausanne
Locations (3):
- Switzerland (3):
  - Lausanne University Hospital (CHUV), Lausanne
  - EHC (Hôpital de Morges), Morges
  - eHnv (Etablissements hospitaliers du nord vaudois), Yverdon-les-Bains

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellet J, Weiss M, Mabire C. Evaluation of a theory-informed implementation of a nursing discharge teaching intervention for older adults. J Adv Nurs. 2023 Aug;79(8):3147-3159. doi: 10.1111/jan.15666. Epub 2023 Apr 4. PMID 37014070
- [Derived] Pellet J, Weiss M, Zuniga F, Mabire C. Implementation and preliminary testing of a theory-guided nursing discharge teaching intervention for adult inpatients aged 50 and over with multimorbidity: a pragmatic feasibility study protocol. Pilot Feasibility Stud. 2021 Mar 17;7(1):71. doi: 10.1186/s40814-021-00812-4. PMID 33731212